CLINICAL TRIAL: NCT06334549
Title: Effects of Vasopressor on Cerebral Oxygenation During General Anesthesia in Abdominal Surgery
Brief Title: A Prospective Study of Vasopressor on Cerebral Oxygenation During General Anesthesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dalian Municipal Central Hospital (Other)
Responsible Party: Principal Investigator, Liping Han, Professor & Vice Director, Dalian Municipal Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSKY2023-107-01
Record Dates: First submitted 2024-03-08; First posted 2024-03-28 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Hypotension Drug-Induced
Keywords: Abdominal surgery; ephedrine; phenylephrine; norepinephrine; cerebral oxygen saturation; MAP; CO; General anesthesia; Propofol; Sevoflurane; Hypotension Drug-induced
MeSH Terms: conditions — Hypotension | interventions — Vasoconstrictor Agents; ephedrine phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Ephedrine-Propofol (Experimental): receive ephedrine 0.15mg/kg (configured concentration 6mg/mL) when MAP was a 20% decrease in baseline blood pressure after both induction of anesthesia and tracheal intubation.
  Interventions: Drug: Ephedrine-P
- Phenylephrine-propofol (Experimental): receive phenylephrine 2.5ug/kg(configured concentration 100ug/mL) when MAP was a 20% decrease in baseline blood pressure after both induction of anesthesia and tracheal intubation.
  Interventions: Drug: Phenylephrine-P
- Norepinephrine-propofol (Experimental): receive norepinephrine 0.2ug/kg(configured concentration 8μg/ml) when MAP was a 20% decrease in baseline blood pressure after both induction of anesthesia and tracheal intubation.
  Interventions: Drug: Norepinephrine-P
- Ephedrine-sevoflurane (Active Comparator): receive Ephedrine 0.15mg/kg(configured concentration 6mg/mL) when MAP was a 20% decrease in baseline blood pressure after both induction of anesthesia and tracheal intubation.
  Interventions: Drug: Ephedrine-S
- Phenylephrine-sevoflurane (Active Comparator): receive phenylephrine 2.5ug/kg(configured concentration 80ug/mL) when MAP was a 20% decrease in baseline blood pressure after both induction of anesthesia and tracheal intubation.
  Interventions: Drug: Phenylephrine-S
- Norepinephrine-sevoflurane (Active Comparator): receive norepinephrine 0.2ug/kg(configured concentration 8ug/mL) when MAP was a 20% decrease in baseline blood pressure after both induction of anesthesia and tracheal intubation.
  Interventions: Drug: Norepinephrine-S

INTERVENTIONS:
Drug: Ephedrine-P — after induction of anesthesia, use total intravenous anesthesia maintained with propofol
  Other Names: vasopressor
  Arms: Ephedrine-Propofol
Drug: Phenylephrine-P — after induction of anesthesia, use total intravenous anesthesia maintained with propofol
  Other Names: vasopressor
  Arms: Phenylephrine-propofol
Drug: Norepinephrine-P — after induction of anesthesia, use total intravenous anesthesia maintained with propofol
  Other Names: vasopressor
  Arms: Norepinephrine-propofol
Drug: Ephedrine-S — after induction of anesthesia, use inhalation anesthesia maintained with sevoflurane
  Other Names: vasopressor
  Arms: Ephedrine-sevoflurane
Drug: Phenylephrine-S — after induction of anesthesia, use inhalation anesthesia maintained with sevoflurane
  Other Names: vasopressor
  Arms: Phenylephrine-sevoflurane
Drug: Norepinephrine-S — after induction of anesthesia, use inhalation anesthesia maintained with sevoflurane
  Other Names: vasopressor
  Arms: Norepinephrine-sevoflurane

SUMMARY:
The purpose of this study is to investigate whether norepinephrine(N), phenylephrine(P) or ephedrine(E) have different effect on cerebral oxygenation in abdominal surgery with propofol or sevoflurane.

DETAILED DESCRIPTION:
This study was a single-center, randomized, double-blinded, controlled trial. First, the effects of E, P, or N on cerebral oxygen saturation(rScO2) under general anesthesia in abdominal surgery were studied. Patients with abdominal surgery were evaluated using near-infrared spectroscopy. Continual changes in systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial blood pressure (MAP), heart rate (HR), stroke volume (SV), cardiac output (CO) and systemic vascular resistance (SVR) will be measured with LiDCO rapidV3 monitoring system. To investigate the individualized therapeutic options & specific mechanisms of the three vasopressors on rScO2 and CO.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III, age 18-80 years
* Elective abdominal surgery
* Signed informed consent

Exclusion Criteria:

* ASA≥IV
* Preoperative unstable blood hemodynamics
* Allergy to ephedrine, phenylephrine or norepinephrine
* Decrease in MAP <20%
* Severe cardiovascular disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Continual changes in Cerebral Oxygen Saturation | 10 minutes after entering the operating room; when 20% decrease in baseline MAP after both induction of anesthesia and intubation; when MAP rising to the highest point after administration of vasopressors
  This outcome is measured by near-infrared spectroscopy

SECONDARY OUTCOMES:
Continual changes in systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial blood pressure (MAP) | 10 minutes after entering the operating room; when 20% decrease in baseline MAP after both induction of anesthesia and intubation; when MAP rising to the highest point after administration of vasopressors
  This outcome is measured by LiDCO rapidV3 monitoring system
Continual changes in heart rate (HR) | 10 minutes after entering the operating room; when 20% decrease in baseline MAP after both induction of anesthesia and intubation; when MAP rising to the highest point after administration of vasopressors
  This outcome is measured by LiDCO rapidV3 monitoring system
Continual changes in stroke volume (SV) | 10 minutes after entering the operating room; when 20% decrease in baseline MAP after both induction of anesthesia and intubation; when MAP rising to the highest point after administration of vasopressors
  This outcome is measured by LiDCO rapidV3 monitoring system
Continual changes in cardiac output (CO) | 10 minutes after entering the operating room; when 20% decrease in baseline MAP after both induction of anesthesia and intubation; when MAP rising to the highest point after administration of vasopressors
  This outcome is measured by LiDCO rapidV3 monitoring system
Continual changes in systemic vascular resistance (SVR) | 10 minutes after entering the operating room; when 20% decrease in baseline MAP after both induction of anesthesia and intubation; when MAP rising to the highest point after administration of vasopressors
  This outcome is measured by LiDCO rapidV3 monitoring system

CONTACTS AND LOCATIONS:
Overall Officials: Hong Fang, MD, Study Chair — Dalian Municipal Central Hospital
Locations (1):
- Dalian Municipal Central Hospital, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No